CLINICAL TRIAL: NCT03065179
Title: Phase II Trial of Stereotactic Body Radiation Therapy in Combination With Nivolumab Plus Ipilimumab in Patients With Metastatic Renal Cell Cancer
Brief Title: SBRT (Stereotactic Body Radiation Therapy) in Combination With Nivolumab/Ipilimumab in Renal Cell Carcinoma (RCC) / Kidney Cancer Patients
Acronym: RADVAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Hans Hammers, Associate Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 072016-044
Record Dates: First submitted 2017-02-07; First posted 2017-02-27 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Kidney Cancer Metastatic; Kidney Cancer; Kidney Cancer, Stage IV
MeSH Terms: conditions — Kidney Neoplasms | interventions — Nivolumab; Ipilimumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab/Ipilimumab plus SBRT (Experimental): Induction Dual Immune Checkpoint Inhibition with nivolumab and ipilimumab plus SBRT to 1-2 metastatic sites, followed by nivolumab monotherapy
  Interventions: Drug: Nivolumab/Ipilimumab; Radiation: SBRT

INTERVENTIONS:
Drug: Nivolumab/Ipilimumab — IV immunotherapy
  Other Names: Opdivo; Yervoy
Radiation: SBRT — SBRT will be delivered in conjunction with immunotherapy
  Other Names: stereotactic radiation

SUMMARY:
This is a multi-institution, single-arm phase II study to determine the safety and efficacy of SBRT (up to 2 metastatic sites preferentially lung, mediastinum or bone in combination of nivolumab and ipilimumab in patients with metastatic renal cell carcinoma(with a clear-cell component and at least 1 measurable metastatic lesion that is not being irradiated).

DETAILED DESCRIPTION:
The study is planned based on a two-stage design that allows early termination for lack of efficacy. A safety run-in phase will be included comprising the first 6 patients at minimum to ensure that the combination of nivolumab plus ipilimumab and SBRT is safe. Then, the investigators will determine whether the combination of nivolumab plus ipilimumab and SBRT yields a clinically compelling antitumor activity measured as objective response rate (ORR), and evaluate other endpoints including Thrombotic thrombocytopenic purpura (TTP), duration of response (DOR), progression free survival (PFS), overall survival (OS) and local control of irradiated sites.

There is no previous experience with SBRT used concurrently with nivolumab and ipilimumab in this study population. Therefore, to ensure that the combination is safe, the first six patients will be treated and observed for toxicity for 6 weeks after radiation before continuing with further accrual. Therefore, six patients will be enrolled at the proposed dose of nivolumab and ipilimumab in combination with SBRT. If 4 out of the first 6 patients experience Grade 3/4 toxicity or a lower grade toxicity requiring immune suppressive therapy during the safety run-in observation period (defined as the first 4-cycles, 12 weeks), enrollment will cease and the study will be halted until further safety analysis of the combination regimen can be performed. If less than 4 out of the first 6 patients experience Grade 3/4 toxicities or require steroids, the investigators will proceed with additional accrual with this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of RCC with a clear-cell component
* Metastatic (AJCC Stage IV) RCC
* Prior adjuvant or neoadjuvant therapy for localized or locally advanced RCC is allowed provided recurrence occurred = or > 6 months after the last dose of the adjuvant or neoadjuvant therapy
* Any number of prior systemic treatment regimen in the advanced/metastatic setting is allowed (cytokine, anti-angiogenic, mammalian target of rapamycin (mTOR) inhibitor or clinical trial) including previously untreated patients
* Karnofsky Performance Status (KPS) of at least 70%
* Life expectancy of at least 3 months
* At least 2 metastatic sites of which at least 1 must be measurable as per RECIST 1.1
* Archival Formalin-fixed paraffin-embedded (FFPE) tumor tissue must be available for correlative studies (Note: Fine Needle Aspiration (FNA) and bone metastases samples are not acceptable for submission)
* Patients with favorable, intermediate and poor risk categories will be eligible for the study. Patients must be categorized according to favorable versus intermediate/poor risk status at registration. International Metastatic RCC Database Consortium (IMDC) must be used to determine prognostic factors

Exclusion Criteria:

* Subjects with previously treated brain or CNS (Central nervous system) metastases are eligible provided that the subject has recovered from any acute effects of radiotherapy and is not requiring steroids, and any whole brain radiation therapy was completed at least 4 weeks prior to study drug administration, or any stereotactic radiosurgery was completed at least 2 weeks prior to study drug administration. Liver metastases will not be included as part of the radiated lesions to be treated.

Medical History and Concurrent Diseases:

* Prior treatment with an anti-Programmed cell death(PD) -1, anti-PD-L1, anti-PD-L2, anti-CD137(cluster of differentiation), or anti-CTLA-4 (cytotoxic T-lymphocyte-associated protein ) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways. Prior treatment with high dose interleukin (HD IL)-2 is allowed.
* Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll. Patients with psoriasis not requiring active, systemic treatment are allowed.
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Uncontrolled adrenal insufficiency
* Requirement for anti-coagulation with Coumadin, low molecular weight heparin and anti-thrombin inhibitors will be accepted if anticoagulation has been stable for at least 4 weeks and no recent history of prior bleeding complications.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast or low risk Gleason 6 prostate cancer
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection
* Known medical condition (eg, a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
* Major surgery (eg, nephrectomy) less than 28 days prior to the first dose of study drug
* Anti-cancer therapy less than 14 days prior to the first dose of study drug or palliative, focal radiation therapy less than 14 days prior to the first dose of study drug
* Presence of any toxicities attributed to prior anti-cancer therapy, other than alopecia, that have not resolved to Grade 1 (NCI CTCAE v4) or baseline before administration of study drug

Physical and Laboratory Test Findings:

* Any of the following laboratory test findings:

  * White blood cell (WBC) < 2,000/mm3
  * Neutrophils < 1,500/mm3
  * Platelets < 100,000/mm3
  * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x ULN (> 5 x ULN if liver metastases are present)
  * Total Bilirubin > 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * Serum creatinine > 1.5 x upper limit of normal (ULN) or creatinine clearance < 40 mL/min (measured or calculated by Cockroft-Gault formula)

Allergies and Adverse Drug Reaction:

* History of severe hypersensitivity reaction to any monoclonal antibody or study drug components

Other Exclusion Criteria:

* Prisoners or subject who are involuntarily incarcerated
* Not suitable for SBRT treatment
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hammers, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 4 participants who signed the informed consent and went through the screening process as part of the protocol and were screen failures.
Period: Overall Study
Arm/Group | Nivolumab/Ipilimumab Plus SBRT
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab/Ipilimumab Plus SBRT
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 57 [35 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events Grade 3 or Higher as Assessed by CTCAE v4.0
Description: An adverse event (AE) will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: up to 35 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab/Ipilimumab Plus SBRT
Number analyzed (Participants) | 25
Participants | 9

2. Primary Outcome: Number of Participants Needing Corticosteroids
Time Frame: up to 35 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab/Ipilimumab Plus SBRT
Number analyzed (Participants) | 25
Participants | 10

3. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as the number of participants with a BOR of CR (Complete response) or PR (Partial response) divided by the number of treated participants. The BOR (Best overall response) is defined as the best response designation, as determined by the investigator, recorded between the date of randomization and the date of objectively documented progression per RECIST 1.1 or the date of first subsequent anti-cancer therapy including radiotherapy, tumor-directed surgery, or systemic anticancer therapy, whichever occurs first. For participants without documented progression or subsequent therapy, all available response designations will contribute to the BOR assessment
Time Frame: up to 35 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab/Ipilimumab Plus SBRT
Number analyzed (Participants) | 25
percentage of participants | 56 [38.7 to 78.9]

ADVERSE EVENTS:
Time Frame: Up to 35 months
Arm/Group | Nivolumab/Ipilimumab Plus SBRT
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab/Ipilimumab Plus SBRT (N=25)
Diarrhea (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
ALT (Alanine Transaminase) (Gastrointestinal disorders) | 1
AST (Aspartate transaminase) (Gastrointestinal disorders) | 1
Amylase (Gastrointestinal disorders) | 6
Lipase (Gastrointestinal disorders) | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab/Ipilimumab Plus SBRT (N=25)
Fatigue (General disorders) | 25
Rash (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Radiation Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 14
Colitis (Gastrointestinal disorders) | 1
ALT (Gastrointestinal disorders) | 3
AST (Gastrointestinal disorders) | 3
Amylase (Gastrointestinal disorders) | 5
Creatinine (Renal and urinary disorders) | 1
Hypothyroidism (Endocrine disorders) | 8
Hyperthyroidism (Endocrine disorders) | 3
Adrenal Insufficiency (Endocrine disorders) | 4
Hypophysitis (Endocrine disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT03065179/Prot_SAP_000.pdf